CLINICAL TRIAL: NCT04856267
Title: Exploration of Arrhythmia Burden in Cardiac Amyloidosis Using Implantable Loop Recorders
Acronym: EXCALIBUR
Status: Completed | Type: Observational
Sponsor: Marianna Fontana (Other)
Responsible Party: Sponsor-Investigator, Marianna Fontana, Professor of Cardiology and Clinical Lead of the UCL Cardiac CMR service, Royal Free Hospital NHS Foundation Trust
Organization: Royal Free Hospital NHS Foundation Trust (Other)
Other Study IDs: 20/NS/0038
Record Dates: First submitted 2021-04-13; First posted 2021-04-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Arrythmia; Cardiac Amyloidosis; Sudden Cardiac Death
Keywords: Implantable Loop Recorder; Arrhythmia; Sudden Cardiac Death; Cardiac Amyloidosis
MeSH Terms: conditions — Arrhythmias, Cardiac; Amyloid Neuropathies, Familial; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Amyloidosis study cohort: Eligible patients will undergo subcutaneous implantation of a cardiac monitor device (Brand name - LINQ device, Medtronic - referred to in the application as "implantable loop recorder" or "ILR")
  Interventions: Device: LINQ device - implantable cardiac monitor - referred to in the application as "implantable loop recorder" or "ILR")

INTERVENTIONS:
Device: LINQ device - implantable cardiac monitor - referred to in the application as "implantable loop recorder" or "ILR") — Implantation of an implantable cardiac monitor device (brand name LINQ device, Medtronic) will be performed under local anaesthetic using an aseptic sterile technique. They will undergo frequent follow-up and monitoring for arrhythmias through remote monitoring of the device

SUMMARY:
The overall aim of this study is to improve our understanding of the effects of the build-up of amyloid deposits in the heart, in particular, our understanding of the risk of abnormal heart beats, or rhythms, associated with people with cardiac (heart) amyloidosis. Symptoms such as palpitations (fast, strong or irregular heart beat) and blackouts are common in people with cardiac amyloidosis, but there is not enough information on what causes this. At present, there is also not enough information on when they occur, how often they happen, and which patients are at risk of having serious, life-threatening types of abnormal heart rhythms.

Some of these abnormal heart rhythms can be treated with medicine; others need electronic devices (e.g. pacemakers) implanted or inserted in the heart to prevent serious harm. The information on when is the best time to implant these life-saving devices remains limited. In this study, a small device known as an implantable loop recorder (ILR) will be implanted under the skin on the chest wall to continuously monitor participants' heart rhythm.

This will help us answer some of the questions about what causes the abnormal heart rhythms, when they happen, and which patients are particularly likely to have them. Furthermore, it may help us to identify earlier, rather than later, those who are at risk of developing abnormal heart rhythms. This may lead to improvements in the care of people with cardiac amyloidosis in the future. Participants may not directly benefit from taking part in this study; however, there is a chance that the ILR may reveal heart rhythm abnormalities in some participants which might not be picked up otherwise, and so may lead to a change in their treatment.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) occurs in up to 1/3 of patients with cardiac amyloidosis but conflicting findings have been reported on the mechanism. Electromechanical dissociation (EMD) is thought to account for some 6-7 cases, underscoring doubts about a role for implantable cardioverter-defibrillators (ICDs). However, there are studies that have described appropriate and effective ICD therapies in 27% to 32% of cases, similar to primary prevention in other disorders. The strength of evidence in all these studies is fairly weak (small, single-centre, retrospective, not linked to mechanism), but this potentially makes ICD implantation more important than in other conditions. It has also been shown in a study with small patient numbers that the pre-terminal event is often bradycardia, which may be amenable to pacemaker therapy. At present, the available information regarding arrhythmia burden in cardiac amyloidosis is limited, and further data are crucial to better guide patient selection for device therapy.

Whilst the burden of arrhythmia and sudden cardiac death appear considerable, there is limited characterisation of the incidence and predictive factors for arrhythmia requiring treatment. Cardiac involvement is the main driver of outcome in cardiac amyloidosis. Amyloidosis is a continuum from small focal amyloid deposits to extensive diffuse myocardial infiltration. The dynamic and progressive nature of amyloid deposition is likely to create an arrhythmogenic substrate that alters over time. For example, patchy amyloid deposits occurring in earlier disease might potentially provide an anatomical substrate enabling re-entry and underlie ventricular tachyarrhythmias, whilst diffuse transmural amyloid deposition may increase risk of AV block and bradyarrythmias. The investigators believe that amyloid deposition will be associated with increased risk of fatal arrhythmias, including AV block, bradyarrhythmias and ventricular arrhythmias. There are no current criteria or arrhythmia risk stratification available to guide device implantation in patients with cardiac amyloidosis. There are also limited data available on predictive disease characteristics that promote arrhythmia

Current monitoring for arrhythmia involves routine 12-lead ECG checks at annual or six-monthly clinic visits. Longer durations of monitoring (24- or 72-hour Holter monitoring or implantable loop recorders, ILR) are undertaken only when clinically indicated. Other cardiac investigations that are routinely performed in cardiac amyloidosis include echocardiography and cardiac magnetic resonance (CMR) imaging.

Current management of arrhythmia is limited to anticoagulation as per the CHADS2VASC score for atrial fibrillation, and permanent pacemaker insertion for standard indications including high degree atrioventricular blocks. There are limited data available to inform insertion of defibrillators, and this is currently assessed on a case by case basis.

Cardiac biomarkers may be helpful in raising clinical suspicion of cardiac amyloidosis patients with known plasma cell dyscrasia and should prompt further investigation with electrocardiogram (ECG) and echocardiography. The combination of cardiac biomarkers serum N-terminal prohormone of brain natriuretic peptide (NT-proBNP) and troponin is useful to stratify prognosis and guide treatment strategies in AL amyloidosis, while NT-proBNP and estimated glomerular filtration rate are used to stratify prognosis in transthyretin amyloid cardiomyopathy (ATTR-CM). In these patients, ECG tends to show low voltage complexes with common observations including repolarisation abnormalities, pseudo-infarction patterns, left anterior hemiblock, ischaemic or non-specific T wave abnormalities, and rhythm disturbances such as atrial fibrillation. Echocardiography shows the cardiac amyloid phenotype is a thick-walled ventricle, small left ventricular chamber volume, valve thickening, atrial enlargement and signs of elevated filling pressures with a restrictive diastolic filling.

CMR is at the forefront of diagnosis and monitoring of cardiac amyloidosis. CMR uses its intrinsic capacity to characterise cardiac tissue on the basis of fundamental MR properties (T1 and T2), and these intrinsic properties can be strengthened by administration of gadolinium-based contrast agents. CMR can visually depict, with late gadolinium enhancement (LGE), and quantify, with T1 mapping, the continuum of cardiac amyloid deposition allowing for noninvasive measurement of cardiac amyloid burden. Transmurality of LGE, elevation in native T1 and extracellular volume fraction (ECV) all correlate with amyloid burden.

In a study from the UK National Amyloidosis Centre (NAC) published in 2015, ILRs were inserted into 20 consecutive patients with severe cardiac AL amyloidosis. The most important finding was that the terminal syncopal phase prior to death revealed initial cardiac decompensation to be associated with marked bradycardia usually caused by complete heart block, subsequently followed by pulseless electrical activity. But this study was done in patients with end stage AL amyloidosis, and rhythm disturbances in the wide spectrum of amyloid infiltration has never been studied.

Currently, arrhythmia risk prediction is limited despite existing structural and functional assessment tools. ILR data would provide invaluable information on arrhythmia burden, which may be correlated with information obtained from the existing standard-of-care (SOC) structural, biochemical and functional assessments such as, but not limited to, T1 mapping and ECV from CMR, serum biomarkers, and the six-minute walk test (6MWT). These data together would provide a global picture of the arrhythmia burden and contributing risk factors; this has the potential to transform our understanding of arrhythmia in cardiac amyloidosis.

Furthermore, improvements in ILR technology have made these devices more patient-friendly. New ILRs no longer require surgical implantation but can be subcutaneously injected in the outpatient setting. They are simple to use, with automatic recording and uploading of data over each 24-hour period for up to 3 years.

An ILR is a small injectable electronic device (approximate size 45 x 7 x 4 mm, about one-third the size of a AAA battery), which is inserted under the skin within the subcutaneous tissue in the chest. It is routinely used for continuous cardiac monitoring for a range of symptoms (syncope, pre-syncope or palpitations of suspected cardiac origin, arrhythmia) in the wider National Health Service (NHS), and at the Royal Free Hospital (RFH). The required incision for device insertion is less than 1 cm, and it can safely be inserted by a trained healthcare professional (HCP) in the outpatient setting. It is safe and well-tolerated once inserted. One suture is required to close the wound.

As with any such procedure there is a small risk of bleeding and/or infection, both of which are rare. The risk of infection may be minimised by the maintenance of aseptic technique and sterile environment throughout the procedure. Patients will remain in the department under observation for 1 hour after the procedure, and the insertion site will be checked for bleeding and any other abnormalities before the patient is allowed to leave.

Patients will attend their GP surgery (or return to the RFH, whichever is their preference) within 7 to 10 days for removal of the suture and for examination of the insertion site. The device may be removed (as per SOC) when the battery runs out or 3 years after insertion, whichever happened first. The device may be removed earlier if indicated by, for example, adverse event. The ILR may also be left in situ once the patient has completed participation or when the battery runs out, according to patient preference.

ILRs are used in routine practice where indicated for continuous cardiac monitoring in patients with later-stage cardiac amyloidosis but are not currently routinely implanted in patients with early stage disease. Although this study will involve implanting ILRs earlier on in the disease process than usual, this is not anticipated to present any additional risk to patients. Therefore the risk categorisation for this trial would be Type A: Comparable to the risk of standard medical care for this particular patient group. Furthermore, there is the potential benefit of early intervention to treat arrhythmias, which could be life-changing and possibly even life-saving for some patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Diagnosed with cardiac AL amyloidosis or cardiac ATTR amyloidosis using standard diagnostic techniques and criteria at the NAC
* Willing and able to provide written informed consent

Exclusion Criteria:

* Patient who already have a cardiac device inserted, such as a permanent pacemaker (PPM), implantable cardioverter-defibrillator (ICD) or implantable cardiac monitor (ILR)
* Other pre-existing cardiac or other pathology which, in the investigators opinion, would adverse affect primary outcome data collection
* Contraindication to CMR imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the National Amyloidosis Centre
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Explore the characteristics (incidence and nature) of significant heart rhythm disturbances in subjects with cardiac amyloidosis by means of implantable cardiac monitor (ILR) | Through study completion, up to 3 years
  Primary outcome measure is the presence of any clinically significant heart rhythm abnormality as revealed from the implantable cardiac monitor (ILR) over the course of the study

SECONDARY OUTCOMES:
Examine the correlation between the characteristics of cardiac arrhythmias, as revealed by implantable cardiac monitor (ILR) with findings from other structural and functional assessment performed as standard of care (SOC) | Through study completion, up to 3 years
  Secondary outcome measure is the correlation of heart rhythm disturbances identified from the implantable cardiac monitor (ILR), with other structural and functional variables obtained from other SOC tests such as, but not limited to, T1 mapping and ECV from CMR, serum biomarkers and the six-minute walk test (6MWT) distance

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Fontana, Principal Investigator — principle investigator
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Falk RH, Comenzo RL, Skinner M. The systemic amyloidoses. N Engl J Med. 1997 Sep 25;337(13):898-909. doi: 10.1056/NEJM199709253371306. No abstract available. PMID 9302305
- [Background] Kyle RA, Gertz MA. Primary systemic amyloidosis: clinical and laboratory features in 474 cases. Semin Hematol. 1995 Jan;32(1):45-59. No abstract available. PMID 7878478
- [Background] Wechalekar AD, Gillmore JD, Hawkins PN. Systemic amyloidosis. Lancet. 2016 Jun 25;387(10038):2641-2654. doi: 10.1016/S0140-6736(15)01274-X. Epub 2015 Dec 21. PMID 26719234
- [Background] Kyle RA, Linos A, Beard CM, Linke RP, Gertz MA, O'Fallon WM, Kurland LT. Incidence and natural history of primary systemic amyloidosis in Olmsted County, Minnesota, 1950 through 1989. Blood. 1992 Apr 1;79(7):1817-22. PMID 1558973
- [Background] Dubrey SW, Cha K, Anderson J, Chamarthi B, Reisinger J, Skinner M, Falk RH. The clinical features of immunoglobulin light-chain (AL) amyloidosis with heart involvement. QJM. 1998 Feb;91(2):141-57. doi: 10.1093/qjmed/91.2.141. PMID 9578896
- [Background] Grogan M, Dispenzieri A. Natural history and therapy of AL cardiac amyloidosis. Heart Fail Rev. 2015 Mar;20(2):155-62. doi: 10.1007/s10741-014-9464-5. PMID 25447844
- [Background] Falk RH, Rubinow A, Cohen AS. Cardiac arrhythmias in systemic amyloidosis: correlation with echocardiographic abnormalities. J Am Coll Cardiol. 1984 Jan;3(1):107-13. doi: 10.1016/s0735-1097(84)80436-2. PMID 6317729
- [Background] Lin G, Dispenzieri A, Kyle R, Grogan M, Brady PA. Implantable cardioverter defibrillators in patients with cardiac amyloidosis. J Cardiovasc Electrophysiol. 2013 Jul;24(7):793-8. doi: 10.1111/jce.12123. Epub 2013 Mar 14. PMID 23489983
- [Background] Varr BC, Zarafshar S, Coakley T, Liedtke M, Lafayette RA, Arai S, Schrier SL, Witteles RM. Implantable cardioverter-defibrillator placement in patients with cardiac amyloidosis. Heart Rhythm. 2014 Jan;11(1):158-62. doi: 10.1016/j.hrthm.2013.10.026. Epub 2013 Oct 10. No abstract available. PMID 24121001
- [Background] Hamon D, Algalarrondo V, Gandjbakhch E, Extramiana F, Marijon E, Elbaz N, Selhane D, Dubois-Rande JL, Teiger E, Plante-Bordeneuve V, Damy T, Lellouche N. Outcome and incidence of appropriate implantable cardioverter-defibrillator therapy in patients with cardiac amyloidosis. Int J Cardiol. 2016 Nov 1;222:562-568. doi: 10.1016/j.ijcard.2016.07.254. Epub 2016 Aug 1. PMID 27513652
- [Background] Epstein AE, Dimarco JP, Ellenbogen KA, Estes NA 3rd, Freedman RA, Gettes LS, Gillinov AM, Gregoratos G, Hammill SC, Hayes DL, Hlatky MA, Newby LK, Page RL, Schoenfeld MH, Silka MJ, Stevenson LW, Sweeney MO; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; American Association for Thoracic Surgery; Society of Thoracic Surgeons. ACC/AHA/HRS 2008 Guidelines for device-based therapy of cardiac rhythm abnormalities. Heart Rhythm. 2008 Jun;5(6):e1-62. doi: 10.1016/j.hrthm.2008.04.014. Epub 2008 May 21. No abstract available. PMID 18534360
- [Background] Andrews CM, Srinivasan NT, Rosmini S, Bulluck H, Orini M, Jenkins S, Pantazis A, McKenna WJ, Moon JC, Lambiase PD, Rudy Y. Electrical and Structural Substrate of Arrhythmogenic Right Ventricular Cardiomyopathy Determined Using Noninvasive Electrocardiographic Imaging and Late Gadolinium Magnetic Resonance Imaging. Circ Arrhythm Electrophysiol. 2017 Jul;10(7):e005105. doi: 10.1161/CIRCEP.116.005105. PMID 28705875
- [Background] Sayed RH, Rogers D, Khan F, Wechalekar AD, Lachmann HJ, Fontana M, Mahmood S, Sachchithanantham S, Patel K, Hawkins PN, Whelan CJ, Gillmore JD. A study of implanted cardiac rhythm recorders in advanced cardiac AL amyloidosis. Eur Heart J. 2015 May 7;36(18):1098-105. doi: 10.1093/eurheartj/ehu506. Epub 2014 Dec 29. PMID 25549725